CLINICAL TRIAL: NCT06122636
Title: Efficacy of a Probiotic and Microbiological Analysis on Oral Complications Induced by Antineoplastic Therapies in Patients With Head and Neck Cancer: Randomized Clinical Study
Brief Title: Efficacy of a Probiotic and Microbiological Analysis on Oral Complications in Patients With HNC
Acronym: HNC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Barcelona (Other)
Responsible Party: Principal Investigator, Tanya Valeria Pereira Riveros, Principal Investigator, University of Barcelona
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 22/2021
Record Dates: First submitted 2023-11-02; First posted 2023-11-08 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Quality of Life; Oral Mucositis; Dental Plaque; Periodontal Diseases; Xerostomia; Dysbiosis
Keywords: Radiotherapy; chemotherapy; surgery; probiotics; head and neck cancer
MeSH Terms: conditions — Stomatitis; Dental Plaque; Periodontal Diseases; Xerostomia; Dysbiosis; Head and Neck Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): An envelope with the same packaging, size, shape and color will be given, it will only differ from the placebo in that it will contain the active ingredient of the intervention which is Lactobacillus Rhamnosus GG, Lactobacillus casei, Streptococcus thermophilus, Bifidobacterium breve, Lactobacillus acidophilus, Bifidobacterium infantis and Lactobacillus bulgaricus.Experimental group
  Interventions: Dietary Supplement: The probiotic to be used in the intervention corresponds to PRODEFEN Plus manufactured by ITALFARMACO S.A. laboratory
- Placebo group (Placebo Comparator): The placebo will be given in an envelope with the same packaging, size, shape and color of contents as the intervention of interest, except that the placebo will not contain the active ingredient of the intervention
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: The probiotic to be used in the intervention corresponds to PRODEFEN Plus manufactured by ITALFARMACO S.A. laboratory — Each patient should take 1 sachet per day, dissolve it in a glass of water, hold in the mouth for 2-3 minutes and then swallow, for a period of 30 days.
  Arms: Experimental group
Other: Placebo — The placebo will be administered in an envelope with the same packaging, size, shape and color of contents as the intervention of interest, except that the placebo will not contain the active ingredient of the intervention.
  Arms: Placebo group

SUMMARY:
The study is a Clinical Trial and the main objective is to Evaluate the effects of probiotics on oral complications induced by antineoplastic therapies in patients with head and neck cancer, attended at the radiotherapy service of the Catalan Institute of Oncology (ICO) Hospitalet and at the Dental Hospital of the University of Barcelona (HOUB), Faculty of Medicine and Health Sciences Bellvitge campus during the period 2022- 2024.

Research question:

Is the use of probiotics compared to placebo effective in reducing oral complications produced by antineoplastic therapies in patients with head and neck cancer attended in the radiotherapy service at the Catalan Institute of Oncology (ICO) Hospitalet and the Dental Hospital of the University of Barcelona, Faculty of Medicine and Health Sciences campus Bellvitge during the period 2022- 2024?

Study population: Patients attended at the radiotherapy service of the Catalan Institute of Oncology (ICO) Hospitalet and at the Dental Hospital of the University of Barcelona (HOUB), (Master of Dentistry in Oncology and Immunocompromised Patients) diagnosed by histological confirmation of head and neck cancer and treated in the last year.Intervention:

Patients who agree to participate in the study will be randomized to the intervention or control group. Two visits will be made, the first as a baseline measurement and the second after the end of the intervention. In the first visit they will be given the products either probiotic or placebo, with presentation of a box with 10 sachets. The probiotics contain: Lactobacillus Rhamnosus GG, Lactobacillus casei, Streptococcus thermophilus, Bifidobacterium breve, Lactobacillus acidophilus, Bifidobacterium infantis and Lactobacillus bulgaricus. 1 x 10e10 Colony Forming Units (CFU). And the placebo composed of excipients. They are gluten free. Each patient will be given 1 sachet dissolved in water, to take 2-3 minutes of mouthfuls then swallow, after brushing, once a day, for 30 days.

DETAILED DESCRIPTION:
Background: The side effects of antineoplastic therapies of the head and neck aggravate the condition of patients resulting in a decrease in the quality of life. At oral level, they can induce the appearance of certain alterations, this predisposes to an imbalance in the oral microbiota, increasing the presence of acidogenic and cariogenic bacteria. In the oral cavity probiotics are associated with a decrease in the colony forming unit (CFU) count of cariogenic pathogens and inhibition of periodontal pathogens. In addition, they modulate the inflammatory response (humoral and cellular). For this reason, they could be considered a good alternative to modulate the oral microbiota in head and neck oncology patients. Hypothesis: The use of probiotics due to the change of the oral microbiota is associated with a beneficial effect against oral complications produced by radiotherapy, chemotherapy and surgery in patients with head and neck cancer, so that probiotic users will have a greater reduction in oral complications induced by cancer therapies compared to those who do not use probiotics. Objectives: To evaluate the effects of probiotics on oral complications induced by antineoplastic therapies in patients with head and neck cancer, attended at the radiotherapy service of the Catalan Institute of Oncology (ICO) Hospitalet and the Dental Hospital of the University of Barcelona (HOUB), Faculty of Medicine and Health Sciences Bellvitge campus during the period 2022- 2024. Methodology: Randomized Clinical Trial during the period 2022-2024. The identification of the population of interest will be patients attended in the radiotherapy service at the Catalan Institute of Oncology (ICO) Hospitalet and at the Dental Hospital of the University of Barcelona (HOUB), in the Master of Dentistry and in Oncology and Immunocompromised Patients. Data will be collected by electronic record, clinical examination, microbiological and radiographic analysis of the participants. Expected results: The use of probiotics is expected to provide a greater reduction in oral complications induced by head and neck antineoplastic therapies. Statistical analysis: Comparison of categorical variables chi-square test, numerical variables Student's test for independent samples and paired samples or Mann-Whitney U test and Wilcoxon signed-rank test. Relative risk with 95% confidence interval. An intention-to-treat analysis will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age.
* Who give informed consent to participate in the study.
* With histologic diagnosis of head and neck cancer.
* Treated within the last year for head and neck cancer.

Exclusion Criteria:

* Patients who do not wish to participate in the study.
* Patients with osteonecrosis.
* Inability to take oral medications.
* Allergic to probiotics.
* On active antibiotic treatment or having received antibiotic treatment in the last thirty days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2022-10-03 (Actual); Primary Completion 2024-12-20 (Actual); Study Completion 2024-12-20 (Actual)

PRIMARY OUTCOMES:
Concentration of oral dysbiosis | 30 days
  Analyzed through microbiological qPCR study with 16 S sRNA primers, real-time quantitative PCR and comparative analysis with conventional culture looking for changes in the total count of the following periodontopathogens: Aggregatibacter actinomycetemcomitans, Porphyromonas gingivalis, Tannerella forsythia, Campylobacter rectus, Fusobacterium nucleatum and Candida culture.
Rate of xerostomia | 30 days
  It will be measured by sialometry, analyzing unstimulated salivary secretion and stimulated salivary secretion
Salivary ph concentration | 30 days
  It will be measured through paper strips, in one of the containers with accumulated saliva.
Rate of oral mucositis | 30 days
  It will be measured through a clinical analysis, taking into account the World Health Organization (WHO) mucositis assessment scale.
Periodontitis rate | 30 days
  Measured by clinical examination according to SEPA (Spanish Society of Periodontology) criteria for the classification of periodontal disease.
Quality of life rate | 30 days
  It will be analyzed based on the quality of life questionnaire for head and neck cancer patients EORTC QLQ-H&N35 Spanish version.

CONTACTS AND LOCATIONS:
Overall Officials: Tanya Pereira Riveros, Msc, Principal Investigator — Universuty of Barcelona
Locations (1):
- University of Barcelona, Barcelona, Spain